CLINICAL TRIAL: NCT07049081
Title: An Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LUCAR-G79 in Subjects With Relapsed/Refractory Autoimmune Diseases (r/r AID)
Brief Title: A Study of LUCAR-G79 in Subjects With Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2404-0001
Record Dates: First submitted 2025-06-20; First posted 2025-07-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Relapsed/Refractory Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor T cells (LUCAR-G79) (Experimental): Each subject will be given a single-dose LUCAR-G79 cells infusion at each dose level.
  Interventions: Biological: LUCAR-G79 T cells

INTERVENTIONS:
Biological: LUCAR-G79 T cells — Prior to infusion of the LUCAR-G79 T cells, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
This is a prospective, single-arm, open-label and dose-escalation Investigator Initialed study to evaluate LUCAR-G79 in adult subjects with relapsed/refractory autoimmune diseases.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LUCAR-G79, a chimeric antigen receptor (CAR) -T cell therapy in subjects with relapsed/refractory autoimmune diseases. Patients who meet the eligibility criteria will receive LUCAR-G79 infusion. The study will include the following sequential stages: screening, pre-treatment (lymphodepleting chemotherapy), treatment (LUCAR-G79 infusion) and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntary agreement to provide written informed consent.
2. Aged 18 to 70 years, either sex.
3. Adequate organ function meet screening criteria.
4. Positive test for cluster of differentiation antigen 19 (CD19).

SLE:

* Have been diagnosed of SLE at least 6 months before screening.
* At screening, antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Smith antibody should be positive.
* Fulfill relapsed/refractory SLE conditions.

SSc:

* Have been diagnosed of SSc before screening.
* At screening, mRSS is higher than 10.
* Fulfill relapsed/refractory SSc conditions.

AAV:

* Have been diagnosed of AAV before screening.
* Antineutrophil Cytoplasmic Antibody (ANCA)-related antibodies meet one of the following conditions: a. Positive for anti-myeloperoxidase (MPO) and/or p-ANCA; b. Positive for anti-proteinase 3 (PR3) and/or c-ANCA.
* Fulfill relapsed/refractory AAV conditions.

IIM:

* Have been diagnosed of IIM before screening.
* Positive test for myositis-associated antibodies or myositis-specific antibodies at screening.
* Fulfill relapsed/refractory IIM conditions.

TAK:

* Have been diagnosed of TAK before screening.
* Active TAK patients meet screening criteria.
* Fulfill relapsed/refractory TAK conditions.

IgG4-RD:

* Have been diagnosed of IgG4-RD before screening.
* Active IgG4-RD patients meet screening criteria.
* Fulfill relapsed/refractory IgG4-RD conditions.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes.
4. Female subjects who were pregnant, breastfeeding.
5. Those with a history of major organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | 2 years after LUCAR-G79 infusion (Day 1)
Incidence of dose-limiting toxicity (DLT) | 2 years after LUCAR-G79 infusion (Day 1)
Pharmacokinetics in peripheral blood | 2 years after LUCAR-G79 infusion (Day 1)
Recommended Dose regimen finding | 2 years after LUCAR-G79 infusion (Day 1)

SECONDARY OUTCOMES:
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 52 weeks for relapsing/refractory systemic lupus erythematosus (r/r SLE) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Change in modified Rodnan skin score (mRSS) from baseline up to 52 weeks for relapsing/refractory systemic sclerosis (r/r SSc) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Change in Birmingham vasculitis activity score (BVAS) from baseline up to 52 weeks for relapsing/refractory anti-neutrophil cytoplastic antibodies (r/r AAV) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Change in manual muscle testing (MMT-8) scores from baseline up to 52 weeks for relapsing/refractory idiopathic inflammatory myopathy (r/r IIM) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Change in Indian Takayasu Activity Score with the Acute-Phase Response (ITAS.A) from baseline up to 52 weeks for relapsing/refractory takayasu arteritis (r/r TAK) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Change in Immune globulin G4-related diseases Response Index (IgG4-RD RI) from baseline up to 52 weeks for relapsing/refractory Immune globulin G4-related diseases (r/r IgG4-RD) subjects | 52 weeks after LUCAR-G79 infusion (Day 1)
Changes from baseline in immunological markers and Immunogenicity (anti-drug antibody) from baseline up to 52 weeks for all subjects | 52 weeks after LUCAR-G79 infusion (Day 1)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Third The People's Hospital of Bengbu, Bengbu, Anhui
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - The second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No